CLINICAL TRIAL: NCT04041414
Title: Feasibility of a Multi-Level School Intervention for LGBTQ Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Jeremy Goldbach, Associate Professor, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1R21MD013971 (NIH)
Record Dates: First submitted 2019-07-03; First posted 2019-08-01 (Actual); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Sexual Minority Stress Experiences Among LGBTQ Youth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention schools (Experimental): Schools will be assigned to either intervention or control schools. Students in intervention schools will receive the intervention in semester 1.
  Interventions: Other: Proud & Empowered!
- Control schools (Active Comparator): Students in control schools will receive no intervention
  Interventions: Other: Proud & Empowered!

INTERVENTIONS:
Other: Proud & Empowered! — Proud & Empowered! is a school-based intervention to decrease sexual minority stress and improve coping among LGBTQ students. It is administered by school counselors and trained social workers.

SUMMARY:
The goal of this R21 grant is to test the feasibility of a theoretically informed, LGBTQ-affirming intervention (Proud & Empowered; P&E). Although LGBTQ adolescents experience disparities in behavioral health outcomes compared to their heterosexual peers, interventions are scarce. For example, LGBTQ adolescents are 3 to 4 times more likely to meet criteria for an internalizing disorder and 2 to 5 times more likely to meet criteria for externalizing disorders than their heterosexual peers. Our intervention seeks to address disparate behavioral health problems such as depression, anxiety and trauma symptomology. Our goal will be achieved by completing two specific aims: 1) Assess the feasibility, including recruitment, enrollment, fidelity of service delivery, satisfaction, safety, and retention, of the intervention in a randomized control trial with four schools, 2) Obtain preliminary estimates of intervention effects on key behavioral health symptoms for LGBTQ youth and school climate (norms, attitudes, beliefs, behaviors) at the school level in preparation for a larger efficacy trial. This innovative R21 application brings together a team of nationally recognized minority stress and prevention science experts and responds to a nationally established public health need for research from the Institute of Medicine, the National Institutes of Health, and the National Gay and Lesbian Task Force.

ELIGIBILITY:
Inclusion Criteria:

* LGBTQ student in one of four high schools

Exclusion Criteria:

* Not meeting inclusion criteria

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - John Muir High School, Pasadena, California
  - Marshall Fundamental High School, Pasadena, California
  - Blair High School, Pasadena, California
  - Pasadena High School, Pasadena, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goldbach JT, Rhoades H, Mamey MR, Senese J, Karys P, Marsiglia FF. Reducing behavioral health symptoms by addressing minority stressors in LGBTQ adolescents: a randomized controlled trial of Proud & Empowered. BMC Public Health. 2021 Dec 23;21(1):2315. doi: 10.1186/s12889-021-12357-5. PMID 34949171

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Schools: Schools will be assigned to either intervention or control schools. Students in intervention schools will receive the intervention in semester 1.
  Proud & Empowered! is a school-based intervention to decrease sexual minority stress and improve coping among LGBTQ students. It is administered by school counselors and trained social workers.
Period: Overall Study
Arm/Group | Intervention Schools | Control Schools
Started | 27 | 20
Completed | 26 | 18
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants who completed the Proud & Empowered intervention. Participants were from four high schools within Los Angeles County. Two schools were assigned to the intervention condition while the other two were assigned to the control condition. Participants were in 9th through 12th grade, and identified as sexual and/or gender minority.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Schools | Control Schools | Total
Number analyzed (Participants) | 26 | 18 | 44
Age, Customized [Count of Participants; unit: Participants]
  13 years | 4 | 0 | 4
  14 years | 4 | 3 | 7
  15 years | 4 | 7 | 11
  16 years | 7 | 5 | 12
  17 years | 6 | 3 | 9
  18 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 6 | 6 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Select all that apply: participants had the option to select multiple responses.
  Participants
    White | 9 | 6 | 15
    Black or African American | 6 | 1 | 7
    Latino or Hispanic | 13 | 10 | 23
    Asian | 2 | 7 | 9
    American Indian or Alaksa Native | 0 | 1 | 1
    Native Hawaiian or Pacific Islander | 0 | 1 | 1
Gender Identity [Count of Participants; unit: Participants]
  Female | 19 | 8 | 27
  Male | 5 | 6 | 11
  Transgender Female | 1 | 0 | 1
  Transgender Male | 1 | 1 | 2
  Genderqueer or gender nonconforming | 0 | 3 | 3
Sexual Orientation [Count of Participants; unit: Participants]
  Gay/Homosexual | 5 | 3 | 8
  Lesbian/Homosexual | 4 | 2 | 6
  Bisexual | 14 | 4 | 18
  Pansexual | 1 | 4 | 5
  Asexual | 1 | 1 | 2
  Queer | 1 | 2 | 3
  Straight/Heterosexual | 0 | 1 | 1
  Decline to Answer | 0 | 1 | 1
Grade in School [Count of Participants; unit: Participants]
  9th Grade | 7 | 1 | 8
  10th Grade | 5 | 8 | 13
  11th Grade | 4 | 5 | 9
  12th Grade | 10 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Sexual Minority Adolescent Stress Inventory (SMASI)
Description: 54-item survey across 10 domains of minority stress. Assesses experiences of minority stress among adolescents. Each statement reflects past-30-day thoughts, feelings, and situations a person may have experienced, with response options of 1 = yes and 0 = no. A total score was calculated by summing the 54 items. The total score ranged from 0-54. Higher values correspond to a worse outcome, meaning the individual in question has had more stressful experiences.
Time Frame: Change between baseline and post-intervention/follow-up (12 weeks).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Schools: Students in intervention schools will receive the intervention in semester 1.
  Proud & Empowered!: Proud & Empowered! is a school-based intervention to decrease sexual minority stress and improve coping among LGBTQ students. It is administered by school counselors and trained social workers.
- Control Schools: Students in control schools will not receive any intervention.
Arm/Group | Intervention Schools | Control Schools
Number analyzed (Participants) | 26 | 18
score on a scale
  Time 1 (Baseline) | 8.44 (6.65) | 7.22 (7.12)
  Time 2 (Post-intervention) | 7.59 (7.13) | 8.29 (7.68)

2. Primary Outcome: Beck Anxiety Inventory (BAI)
Description: 21-item self-report assessment of anxiety symptoms. The total score is calculated by taking the sum of the 21 items. There are five responses an individual can choose from for each item, these being "Not at all" which is scored as a 1, "Mildly, but it didn't bother me much" which is scored as a 2, "Moderately -- It wasn't pleasant at times" which is scored as a 3, "Severely -- It bothered me a lot" which is scored as a 4, and "Decline to answer" which is scored as a 5. The total score ranges from 0-63. Higher values indicate higher self-reported anxiety: Score of 0-21 indicates low anxiety, Score of 22-35 indicates moderate anxiety, Scores of 36+ indicates potentially concerning levels of anxiety. Subscales are calculated through summation.
Time Frame: Change between baseline and post-intervention/follow-up (12 weeks).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Schools | Control Schools
Number analyzed (Participants) | 26 | 18
score on a scale
  Time 1 (Baseline) | 22.08 (14.44) | 26.89 (16.75)
  Time 2 (Post-intervention) | 19.56 (16.08) | 27.39 (14.14)

3. Primary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: 20-item self-report assessment of post-traumatic stress disorder (PTSD) symptoms which addresses all 20 DSM-5 symptoms of PTSD. A total symptom severity score can be calculated by summing the scores for each of the 20 items. Each item has five possible responses including "Not at all" which is scored as a 0, "A little bit" which is scored as a 1, "Moderately" which is scored as 2, "Quite a bit" which is scored as a 3, and "Extremely" which is scored as a 4. The potential range of scores is 0-80. Higher scores indicate a worse outcome where the individual has higher severity of PTSD symptoms.
Time Frame: Change between baseline and post-intervention/follow-up (12 weeks).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Schools | Control Schools
Number analyzed (Participants) | 26 | 18
score on a scale
  Time 1 (Baseline) | 21.81 (18.30) | 26.78 (20.34)
  Time 2 (Post-intervention) | 24.40 (19.08) | 29.28 (17.32)

4. Primary Outcome: Beck Depression Inventory
Description: 21-item self-report assessment of depression symptoms and severity of depression. The items are rated on a 4-point scale ranging from 0-3 based on the severity of each item (e.g., 0=I do not feel sad, 1=I feel sad much of the time, 2=I am sad all the time, and 3=I am so sad or unhappy that I can't stand it). The total range of scores is from 0-63. Higher values indicate a worse outcome and indicates a greater severity of depression. Scores of 0-13 indicates minimal depression, scores of 14-19 indicates mild depression, scores of 20-28 indicates moderate depression, scores of 29-63 indicates severe depression. Subscale values are achieved through summation.
Time Frame: Change between baseline and post-intervention/follow-up (12 weeks).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Schools | Control Schools
Number analyzed (Participants) | 26 | 18
score on a scale
  Time 1 (Baseline) | 15.40 (11.54) | 17.81 (9.56)
  Time 2 (Post-intervention) | 15.68 (11.96) | 18.65 (12.77)

5. Primary Outcome: Coping Strategies Inventory
Description: 16-item assessment measuring specific coping strategies people use in response to stressful events. Individuals respond to 16 items, with each item assessing components of Problem Solving, Cognitive Restructuring, Social Support, Express Emotions, Problem Avoidance, Wishful Thinking, and Social Withdrawal. Individuals can respond in 5 different ways, these being "Never", "Seldom", "Sometimes", "Often", or "Almost Always". These responses are scored from 1-5 with "Never" being a 1 and "Almost Always" being a 5. The total score is a summation of item scores with a range from 16-80. Higher scores in a particular primary scale indicates that the individual implements that form of coping strategy more often.
Time Frame: Change between baseline and post-intervention/follow-up (12 weeks).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Schools | Control Schools
Number analyzed (Participants) | 26 | 18
score on a scale
  Time 1 (Baseline) | 49.96 (15.23) | 47.85 (12.48)
  Time 2 (Post-intervention) | 47.64 (16.25) | 49.26 (14.22)

6. Primary Outcome: Adapted CSSRS Suicide Questions (Columbia Suicide Severity Rating Scale)
Description: Six items assessing current suicidality that were adapted from the longer, treatment-based Columbia Suicide Severity Rating Scale. The first two items ask about passive ideation and active ideation, and affirmative responses link to follow-up questions about methods, intent, plans, and attempts. The scale is scored as follows: 0 = no to passive ideation and no to active ideation
  1. = yes to passive ideation (but no to active ideation)
  2. = yes to active ideation (but no method, intent, plan)
  3. = yes to method (but no intent or plan)
  4. = yes to intent (but no plan)
  5. = yes to plan Attempts can be scored on its own or added to the overall scale for a risk score of 6 if participant has a recent suicide attempt.
Time Frame: Change between baseline and post-intervention/follow-up (12 weeks).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Schools | Control Schools
Number analyzed (Participants) | 26 | 18
score on a scale
  Time 1 (Baseline) | 0.63 (1.31) | 0.5 (1.34)
  Time 2 (Post-intervention) | .71 (1.46) | 0.61 (1.24)

7. Secondary Outcome: Youth Risk Behavior Survey Substance Use Questions
Description: Measures individual's usage of various substances in their lifetime and within the past 30 days as well as the ways in which individuals have used marijuana, tobacco, or nicotine in the past 30 days. Each substance is individually analyzed for both lifetime usage and past 30 day usage. Individuals can answer Yes or No for both lifetime usage and past 30 day usage. Each substance can range from 0 to the maximum number of survey responses. In addition, for marijuana, students can specify the way in which they used it with response options of smoking, vaping, edible or beverage form, or other. For nicotine and tobacco, students can specify the way in which they used it with the response options of smoking, vaping, or other. "Yes" responses indicate a worse outcome indicating that individuals have used or are currently using the substance in question.
Time Frame: Change between baseline and post-intervention/follow-up (12 weeks).
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Intervention Schools | Control Schools
Number analyzed (Participants) | 26 | 18
participants
  Alcohol Use : Time 1 (Baseline) | 11 | 5
  Alcohol Use : Time 2 (Post-intervention) | 12 | 7
  Tobacco Use : Time 1 (Baseline) | 6 | 2
  Tobacco Use : Time 2 (Post-intervention) | 5 | 4
  Marijuana Use : Time 1 (Baseline) | 9 | 0
  Marijuana Use : Time 2 (Post-intervention) | 10 | 1
  Pain Relievers Use : Time 1 (Baseline) | 3 | 1
  Pain Relievers Use : Time 2 (Post-intervention) | 1 | 1
  Tranquilizers Use : Time 1 (Baseline) | 0 | 0
  Tranquilizers Use : Time 2 (Post-intervention) | 0 | 0
  Stimulants Use : Time 1 (Baseline) | 0 | 0
  Stimulants Use : Time 2 (Post-intervention) | 1 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks, from pre-test to post-test.
Arm/Group | Intervention Schools | Control Schools
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/20
Other Adverse Events (participants affected / at risk) | 0/27 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT04041414/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT04041414/ICF_001.pdf